CLINICAL TRIAL: NCT06589297
Title: Prognostic Value for Predicting Functional Outcome Bioimpedancemetry and Temporal Muscle Measurement in Acute Stroke
Brief Title: Body Composition and Acute Stroke
Acronym: PREDISTROKE
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Régional d'Orléans (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: CHUO-2024-04
Record Dates: First submitted 2024-09-03; First posted 2024-09-19 (Actual); Last update posted 2026-02-02 (Actual); Status verified 2026-01

CONDITIONS: Acute Stroke
Keywords: Stroke; Body composition; Bioimpedancemetry; Temporal muscle; Sarcopenia
MeSH Terms: conditions — Stroke; Sarcopenia

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Acute stroke patients (Other): Acute stroke patients
  Interventions: Diagnostic Test: Modified Rankin scale

INTERVENTIONS:
Diagnostic Test: Modified Rankin scale — Acute stroke patients will undergo modified rankin scale

SUMMARY:
Body composition appears to be a prognostic factor for the severity and functional outcome of stroke patients. In this study the prognostic value of two bioimpedance parameters will be studied (skeletal mass index and phase angle) and two temporal muscle measurements (thickness and surface area) to predict the functional outcome of patients at discharge and at 6 months

DETAILED DESCRIPTION:
A stroke commonly causes weakness and loss of independence. Predicting functional outcomes is a major challenge because it guides rehabilitation care or institutionalization choices. Various factors, including the extent of the initial deficit or the size of the lesion, have been shown to play a role in residual disability after stroke. Premorbid physiological status has been less studied in stroke. However, loss of muscle mass and premorbid strength are prognostic factors for poor short- and medium-term functional recovery.

In this work, the body composition of patients in the acute phase of a stroke will be studied to determine whether its alteration is a poor prognostic factor in the short term (discharge from the initial hospitalization) and in the medium term (follow-up visit at 6 months). It will be studied using impedance analysis and morphological measurements on the temporal muscle.

In a cohort study of hospitalized patients in the acute phase of a stroke, measurements using a bioimpedance meter (InBody BWA) will be performed to measure a skeletal mass index (SMI) and phase angle. The properties of the temporal muscle (thickness and surface) will also be measured at T1, within 72 first hours after the stroke. Clinical and morphological data will also be collected (weight, height, initial deficit, lesion volume).

The aim of the work is to determine whether these body composition factors have an impact on the functional outcome of patients assessed at discharge and 6 months later. Functional assessment will be performed with modified Rankin score (mRS).

It is hypothesized that all body composition factors studied will be factors independent of the short- and medium-term functional prognosis.

ELIGIBILITY:
Inclusion Criteria:

* volunteer stroke patients in acute phase
* Age ≥ 18 years
* Having had a brain MRI
* Able to understand assessment guidelines
* Not having objected to participate in the study after being duly informed

Exclusion Criteria:

* Person under tutorship or curatorship
* Person under court protection
* Persons deprived of their liberty
* Pregnant or breastfeeding women
* Have a pacemaker or defibrillator

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 250 (Estimated)
Dates: Start 2024-10-10 (Actual); Primary Completion 2028-06 (Estimated); Study Completion 2028-06 (Estimated)

PRIMARY OUTCOMES:
phase angle | 72 hours after stroke
thickness of temporal muscle | 72 hours after stroke
surface area of temporal muscle | 72 hours after stroke

SECONDARY OUTCOMES:
Modified Rankin Scale (mRS) | Month 6
  The modified Rankin Scale is used to assess the disability of patients in the acute phase of stroke recovery. It consists of a single item, with 5 levels corresponding to no disability, mild disability, moderate disability, moderately severe disability and severe disability.
Modified Rankin Scale (mRS) | Through month 3
  The modified Rankin Scale is used to assess the disability of patients in the acute phase of stroke recovery. It consists of a single item, with 5 levels corresponding to no disability, mild disability, moderate disability, moderately severe disability and severe disability.
skeletal muscular Index | 72 hours after stroke

CONTACTS AND LOCATIONS:
Overall Officials: Marc VERIN, PUPH, Principal Investigator — CHU ORLEANS
Locations (1):
- CHU d'ORLEANS, Orléans, France

REFERENCES:
- [Background] Amir A, Pittel Z, Shahar A, Fisher A, Heldman E. Cholinotoxicity of the ethylcholine aziridinium ion in primary cultures from rat central nervous system. Brain Res. 1988 Jun 28;454(1-2):298-307. doi: 10.1016/0006-8993(88)90830-x. PMID 3409012
- [Background] Nozoe M, Kubo H, Kanai M, Yamamoto M, Okakita M, Suzuki H, Shimada S, Mase K. Reliability and validity of measuring temporal muscle thickness as the evaluation of sarcopenia risk and the relationship with functional outcome in older patients with acute stroke. Clin Neurol Neurosurg. 2021 Feb;201:106444. doi: 10.1016/j.clineuro.2020.106444. Epub 2021 Jan 1. PMID 33395619
- [Background] Katsuki M, Kakizawa Y, Nishikawa A, Yamamoto Y, Uchiyama T, Agata M, Wada N, Kawamura S, Koh A. Temporal Muscle and Stroke-A Narrative Review on Current Meaning and Clinical Applications of Temporal Muscle Thickness, Area, and Volume. Nutrients. 2022 Feb 6;14(3):687. doi: 10.3390/nu14030687. PMID 35277046
- [Background] Li YX, Hou J, Liu WY. Long-term prognostic significance of sarcopenia in acute ischemic stroke. Medicine (Baltimore). 2022 Aug 26;101(34):e30031. doi: 10.1097/MD.0000000000030031. PMID 36042682
- [Background] Nagano A, Shimizu A, Maeda K, Ueshima J, Inoue T, Murotani K, Ishida Y, Mori N. Predictive Value of Temporal Muscle Thickness for Sarcopenia after Acute Stroke in Older Patients. Nutrients. 2022 Nov 27;14(23):5048. doi: 10.3390/nu14235048. PMID 36501078
- [Background] Dubinski D, Won SY, Mattes I, Trnovec S, Behmanesh B, Cantre D, Baumgarten P, Dinc N, Konczalla J, Wittstock M, Freiman TM, Gessler F. Frailty in cerebellar ischemic stroke-The significance of temporal muscle thickness. Front Neurol. 2023 Sep 26;14:1193685. doi: 10.3389/fneur.2023.1193685. eCollection 2023. PMID 37822528
- [Background] Namgung HG, Hong S, Choi YA. Association of Temporalis Muscle Mass with Early Cognitive Impairment in Older Patients with Acute Ischemic Stroke. J Clin Med. 2023 Jun 15;12(12):4071. doi: 10.3390/jcm12124071. PMID 37373767